CLINICAL TRIAL: NCT00415506
Title: A PhaseI/II Prospective, Randomized, Dose-Ranging Pilot Study of Rituximab in the Treatment of Refractory Scleritis and Non-Infectious Orbital Inflammation
Brief Title: Rituximab in the Treatment of Scleritis and Non-Infectious Orbital Inflammation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Jim Rosenbaum, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: e1529
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Scleritis; Orbital Disease
MeSH Terms: conditions — Scleritis; Orbital Diseases | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Scleritis (Experimental): Subjects with Scleritis
  Interventions: Drug: Rituximab
- Orbital Inflammation (Experimental): Subjects with Orbital Inflammation
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Two 500 or 1000mg infusions over 2 weeks with the option of retreating after 6 months if initial improvement was seen.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of Rituximab in refractory scleritis and non-infectious orbital inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-infectious scleritis or idiopathic orbital inflammatory disease requiring chronic immunosuppressive treatment for disease control.
* Intolerance, failure to respond to, or inability to taper below prednisone > 10mg/day in addition to one systemic immunosuppressive (such as methotrexate, azathioprine, mycophenolate mofetil, cyclosporine, cyclophosphamide, or chlorambucil).
* Patients must be on a stable dosage of prednisone and at least one steroid-sparing agent in the 30 days prior to screening/enrollment.
* Active disease will be defined using physician judgment and supported by patient and physician global ocular disease assessment of > 5 cm on a 10cm visual analog scale anchored by the words "Inactive Eye Disease" at 0 cm point and "Extremely Active Eye Disease" at the 10cm point. Investigator discretion may apply in some cases.
* Selected patients who are on biological agents such as TNF blockers etanercept, infliximab and adalimumab with ongoing ocular disease are acceptable. There will be an 8 week washout period of etanercept and a 12 week washout period for infliximab and adalimumab before patients are dosed with rituximab.
* In patients with concomitant systemic autoimmune diseases including RA, SLE, Sjogrens, Wegener's granulomatosis the systemic disease must be sufficiently stable and not life threatening to allow tapering of steroids and/or immunosuppressive agents thus allowing assessment of ocular effect of rituximab.
* Adults of both genders > 18 years old. There is no upper age limit as long as there are no other disqualifying health conditions.
* Have had a recent (<3 months old) PPD skin test and are considered eligible according to the tuberculosis (TB) screening, eligibility assessment, and prevention rules defined in Appendix C.
* Screening laboratory test results should be acceptable to the Investigator prior to placing a patient on study drug.
* Must have a chest radiograph within 3 months prior to first infusion with no evidence of malignancy, infection or fibrosis.
* Adequate renal function as indicated by normal BUN and creatinine levels.

Exclusion Criteria:

* Untreated thyroid disease
* Organ threatening systemic disease as evidenced by rapidly progressive glomerulonephritis, pulmonary hemorrhage or respiratory failure, seizures or psychosis, progressive neuropathy or myopathy

General Safety & Laboratory Exclusion Criteria

Patients will be excluded from the study based on the following criteria:

* Hemoglobin: < 8.5 gm/dL
* Platelets: < 100,000/mm
* AST or ALT >2.5 x Upper Limit of Normal unless related to primary disease.
* Positive Hepatitis B or C serology (Hep B Surface antigen and Hep C antibody)
* History of positive HIV (HIV conducted during screening if applicable)
* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 4 weeks prior to randomization
* Previous Treatment with Rituximab (MabThera® / Rituxan®)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of recurrent significant infection or history of recurrent bacterial infections
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening, or oral antibiotics within 2 weeks prior to screening
* Unstable steroid dose in the past 4 weeks
* Lack of peripheral venous access
* History of drug, alcohol, or chemical abuse within 6 months prior to screening
* Pregnancy (a negative serum pregnancy for all women of childbearing potential at screening and negative urine pregnancy test prior to each infusion) or lactation
* Concomitant or previous malignancies, with the exception of curatively resected non-melanoma skin carcinomas or carcinoma in situ of the cervix
* History of psychiatric disorder that would interfere with normal participation in this protocol
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Inability to comply with study and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James T Rosenbaum, MD, Principal Investigator — Oregon Health and Science University; Eric B Suhler, MD, Study Director — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Suhler EB, Lim LL, Beardsley RM, Giles TR, Pasadhika S, Lee ST, de Saint Sardos A, Butler NJ, Smith JR, Rosenbaum JT. Rituximab therapy for refractory orbital inflammation: results of a phase 1/2, dose-ranging, randomized clinical trial. JAMA Ophthalmol. 2014 May;132(5):572-8. doi: 10.1001/jamaophthalmol.2013.8179. PMID 24652467

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from January 2007 through March of 2010. Subjects were recruited from the investigator's medical clinic.
Pre-assignment Details: Of the 20 subjects enrolled, two subjects had both orbital disease and scleritis. These two subjects were followed for both indications.
Groups:
- Scleritis: Patients with non-infectious scleritis and is a phase II, randomized, double-blinded, prospective clinical trial of two different doses of rituximab to compare the safety and efficacy of these 2 doses. Patients will be randomized to either 500 mg or 1000 mg of rituximab administered intravenously two weeks apart.
- Orbital Inflammation: Patients with non-infectious orbital inflammatory disease, and is a phase I, prospective clinical trial to examine the safety of the 2 infusions of rituximab intravenously, 2 weeks apart, in the treatment of non-infectious orbital inflammation. The first 5 patients will receive 1000 mg of rituximab at each infusion, any additional patients will be randomized to receive either 500 mg or 1000 mg of rituximab.
Period: Overall Study
Arm/Group | Scleritis | Orbital Inflammation
Started | 12 | 10
Completed | 9 | 9
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scleritis | Orbital Inflammation | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 8 | 20
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Medications
Description: Reduction (decrease in dosage) of systemic corticosteroids or immunosuppressive therapy by at least 50% by 24 weeks.
Time Frame: 24 Weeks
Population: Only patients currently on systemic corticosteroids were analyzed for this outcome point.
Measure: Number; unit: participants
Arm/Group | Scleritis | Orbital Inflammation
Number analyzed (Participants) | 11 | 6
participants | 5 | 4

2. Primary Outcome: Improved Control of Inflammation
Description: For patients with scleritis, disease activity as measured by a modified grading system first described by McCluskey et al. (McCluskey and Wakefield 1987; McCluskey and Wakefield 1991). Improvement in scleritis activity will be defined as a reduction in this grading score of 2 or more, or an overall score of 4 or less by 24 weeks.
  For patients with orbital inflammation, disease activity as measured by a modified grading system first devised by Werner (Werner 1977). Improvement in orbital inflammation will be defined as a reduction in this grading score of 2 or more, or an overall score of 3 or less.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Scleritis | Orbital Inflammation
Number analyzed (Participants) | 12 | 10
participants | 9 | 7

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each subject during study participation, up to 48 weeks.
Arm/Group | Orbital Inflammation | Scleritis
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes